CLINICAL TRIAL: NCT00753467
Title: Protocol Title: A Phase II Open-labeled Study to Determine the Safety and Preliminary Efficacy of Interferon-gamma 1b (IFN-γ 1b) in Patients With Chronic Hepatitis B Who Are HBV DNA Positive
Brief Title: A Phase II Study to Determine the Safety and Efficacy of Interferon-gamma in Patients With Chronic Hepatitis B
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Huntington Medical Research Institutes (Other)
Collaborators: InterMune (Industry)
Responsible Party: Myron Tong, PhD, MD, HMRI
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TONG-HBV-0801
Record Dates: First submitted 2008-09-15; First posted 2008-09-16 (Estimated); Last update posted 2010-10-21 (Estimated); Status verified 2008-09

CONDITIONS: Hepatitis B
Keywords: HBV; Treatment; Interferon-gamma; combination; Hepsera; Actimmune; HBV DNA
MeSH Terms: conditions — Hepatitis B | interventions — interferon gamma-1b; Interferon-gamma; adefovir dipivoxil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Experimental): IFN-γ 1b monotherapy: 200 micro-grams daily for 30 days
  Interventions: Drug: IFN-γ 1b (Actimmune)
- 2 (Experimental): IFN-γ 1b 200 micro-grams daily) combination therapy with Adefovir dipivoxil (10 mg daily) for 30 days
  Interventions: Drug: IFN-γ 1b and Adefovir dipivoxil combination
- 3 (Active Comparator): Adefovir dipivoxil monotherapy (10 mg QD) 30 days
  Interventions: Drug: Adefovir dipivoxil

INTERVENTIONS:
Drug: IFN-γ 1b (Actimmune) — IFN-γ 1b: 200μg given SC ED = 2 vials of active drug (0.5 mL from each vial) will be mixed for a total volume of 1.0 mL per dose
  Other Names: Interferon gamma; Actimmune; Immune Interferon; IFN-gamma
  Arms: 1
Drug: Adefovir dipivoxil — Adefovir dipivoxil: 1 tablet of 10mg given orally QD
  Other Names: Hepsera
  Arms: 3
Drug: IFN-γ 1b and Adefovir dipivoxil combination — IFN-γ 1b: 200μg given SC ED = 2 vials of active drug (0.5 mL from each vial) will be mixed for a total volume of 1.0 mL per dose Adefovir dipivoxil: 1 tablet of 10mg given orally QD
  Other Names: Actimmune; Interferon gamma; IFN gamma; Immune Interferon; Hepsera
  Arms: 2

SUMMARY:
Open-label, prospective, two part study evaluating IFN-γ 1b at a dose of 200μg by subcutaneous injection every day either alone or in combination with Adefovir dipivoxil or Adefovir dipivoxil alone at a dose of 10mg QD in patients with chronic Hepatitis B.

DETAILED DESCRIPTION:
After signing the informed consent potential patients will undergo a screening medical history, physical examination, and laboratory tests.

The study will consist of two parts:

* Part A: IFN-γ 1b monotherapy
* Part B: IFN-γ 1b combination therapy with Adefovir dipivoxil or Adefovir dipivoxil monotherapy

Patients will be enrolled sequentially into to one of three treatment groups. In Part A, ten patients will be enrolled and will receive IFN-γ 1b 200μg, administered every day by subcutaneous injection for 4 weeks. If HBV DNA is reduced by ≥ 1 log10 copies/ mL in ≥ 30% of patients the protocol will proceed to Part B.

In Part B, twenty patients will be enrolled into two cohorts (total of 10 for each cohort) and treated for four weeks. The two cohorts will be administered:

* IFN-γ 1b 200μg, administered every day combination therapy with Adefovir dipivoxil (10mg QD) or
* Adefovir dipivoxil (10mg QD) alone

On the initial study visit, patients will be given instruction on self injection of IFN-γ 1b (if applicable). Patients will be monitored for safety, tolerability, HBV DNA, clinical chemistries including a standard panel of liver tests and hematologies throughout the study and for the two week post-treatment observation period.

ELIGIBILITY:
Inclusion Criteria:

Patients must fulfill all of the following criteria to be eligible for enrollment into the study:

1. Men or women age 18 to 75 years
2. Chronic hepatitis B infection based on a history of positive anti-HBsAg and positive for HBV DNA and with or without elevations in liver tests (test to be repeated on screening)

Exclusion Criteria:

Patients with any of the following will be excluded from randomization:

1. Presence of clinically evident cirrhosis including: ascites requiring active diuretic therapy, history of or therapy for hepatic encephalopathy, or history of GI variceal bleeding
2. Platelet count < 50,000/mm3
3. Serum ALT level > 10 times upper limit of normal
4. Alpha-fetoprotein level ≥ 200 ng/mL or alpha-fetoprotein level between 50-200 ng/mL in association with liver ultrasound or other radiographic abnormality suspicious for hepatic neoplasm
5. Serum creatinine level > 1.6 mg/dL
6. Hematology outside of specified limits: neutrophil count <1000/mm3, hemoglobin <10 g/dL in males and <9 g/dL in females
7. Unstable or uncontrolled thyroid disease
8. Treatment with any interferon-α or nucleoside/tide analog within the previous 4 weeks
9. Presence of clinically significant cryoglobulinemia (e.g., skin rash, arthritis, or renal insufficiency due to cryoglobuliemia)
10. Presence or history of autoimmune hepatitis, alpha-1 anti-trypsin deficiency, hemochromatosis, Wilson's disease, drug- or toxin-induced liver disease, alcohol-related liver disease, primary biliary cirrhosis, or sclerosing cholangitis (mild-to-moderate steatosis is acceptable)
11. Chronic hepatitis C infection
12. Hepatits Delta infection (HDV)
13. Known history of HIV infection or positive HIV antibody test by Western Blot (test performed within 60 days of screening can be used to determine eligibility)
14. A disease known to cause significant alteration in immunologic function including hematological malignancy or autoimmune disorder (e.g. rheumatoid arthritis, systemic lupus erythematosis, autoimmune thyroid disease, leukemia, lymphoma, etc)
15. Concurrent therapy with immunosuppressive drugs or cytotoxic agents such as oral prednisone, cyclosporine, azathioprine, or chemotherapeutic agent(s) (e.g., cyclophosphamide, methotrexate, or cancer chemotherapy) or radiation therapy
16. Behavior that suggests a significant risk of poor compliance including, but not limited to:

    1. Illicit drug abuse within the past 3 years
    2. Current or history of alcohol abuse within the past 2 years
17. Prior treatment with IFN-γ 1b
18. History of unstable or deteriorating cardiac disease, including but not limited to:

    1. Myocardial infarction, coronary artery bypass surgery, or angioplasty within the past 6 months
    2. Congestive heart failure requiring hospitalization within the past 6 months
    3. Uncontrolled arrhythmias
    4. Transient ischemic attacks (TIAs)
    5. Any cardiac condition that, in the opinion of the site PI, might be significantly exacerbated by flu-like symptoms associated with the administration of IFN γ 1b
19. Preexisting (within last two years) or active psychiatric condition including severe depression, major psychoses, suicidal ideation or suicidal attempts
20. History of (within last two years) or current neurologic or psychiatric disorder that, in the opinion of the site PI, might be exacerbated by flu-like symptoms associated with the administration of IFN γ 1b. In addition, patients with the following conditions should be excluded:

    1. History of multiple sclerosis
    2. Seizures within the past 2 years
21. Severe or poorly controlled diabetes
22. Pregnancy or lactation. Females of childbearing potential are required to have a negative urine pregnancy test prior to treatment and must agree to practice abstinence or prevent pregnancy by at least a barrier method of birth control for the duration of the study
23. Hemoglobinopthies (e.g. thalassemia, sickle cell disease)
24. Any serious or chronic disease that, in the opinion of the Principal Investigator (PI), may affect the assessment of safety or efficacy parameters. This includes, but is not limited to, patients with malignancy who are receiving chemotherapy, chronic obstructive pulmonary disease or asthma requiring maintenance oral steroids, or active kidney disease
25. Any condition which, in the opinion of the site PI, is likely to result in the death of the patient within the next year
26. Patients who, in the opinion of the site PI, are not suitable candidates for enrollment or would not comply with the requirements of the study
27. Patients who have had a liver transplant
28. Patients who have Adefovir mutations on baseline tests

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2008-09; Primary Completion 2009-08 (Estimated); Study Completion 2009-08 (Estimated)

PRIMARY OUTCOMES:
The primary objective is to evaluate the safety and tolerability of IFN-γ 1b either alone or in combination with Adefovir dipivoxil in patients with chronic Hepatitis B. | 30 days

SECONDARY OUTCOMES:
Evaluate the changes in serum HBV DNA concentrations following administration of Adefovir dipivoxil alone, IFN-γ 1b either alone or in combination with Adefovir dipivoxil in patients with chronic Hepatitis B. | 30 days
Evaluate the changes in liver tests and hematology following administration of Adefovir dipivoxil alone, IFN-γ 1b either alone or in combination with Adefovir dipivoxil in patients with chronic Hepatitis B. | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Myron J Tong, Phd, MD, Study Chair — HMRI
Locations (1):
- Huntington Medical Research Institutes, Pasadena, California, United States

REFERENCES:
- [Background] Parvez MK, Sehgal D, Sarin SK, Basir SF, Jameel S. Inhibition of hepatitis B virus DNA replicative intermediate forms by recombinant interferon-gamma. World J Gastroenterol. 2006 May 21;12(19):3006-14. doi: 10.3748/wjg.v12.i19.3006. PMID 16718779
- [Background] Lau JY, Lai CL, Wu PC, Chung HT, Lok AS, Lin HJ. A randomised controlled trial of recombinant interferon-gamma in Chinese patients with chronic hepatitis B virus infection. J Med Virol. 1991 Jul;34(3):184-7. doi: 10.1002/jmv.1890340310. PMID 1919540
- [Background] Marcellin P, Loriot MA, Boyer N, Martinot-Peignoux M, Degott C, Degos F, Brandely M, Lenfant B, Benhamou JP. Recombinant human gamma-interferon in patients with chronic active hepatitis B: pharmacokinetics, tolerance and biological effects. Hepatology. 1990 Jul;12(1):155-8. doi: 10.1002/hep.1840120124. PMID 2115494
- [Result] Narayan R, Buronfosse T, Schultz U, Chevallier-Gueyron P, Guerret S, Chevallier M, Saade F, Ndeboko B, Trepo C, Zoulim F, Cova L. Rise in gamma interferon expression during resolution of duck hepatitis B virus infection. J Gen Virol. 2006 Nov;87(Pt 11):3225-3232. doi: 10.1099/vir.0.82170-0. PMID 17030856
- [Result] Wang J, Michalak TI. Inhibition by woodchuck hepatitis virus of class I major histocompatibility complex presentation on hepatocytes is mediated by virus envelope pre-S2 protein and can be reversed by treatment with gamma interferon. J Virol. 2006 Sep;80(17):8541-53. doi: 10.1128/JVI.00830-06. PMID 16912304
- [Result] Wieland SF, Eustaquio A, Whitten-Bauer C, Boyd B, Chisari FV. Interferon prevents formation of replication-competent hepatitis B virus RNA-containing nucleocapsids. Proc Natl Acad Sci U S A. 2005 Jul 12;102(28):9913-7. doi: 10.1073/pnas.0504273102. Epub 2005 Jul 1. PMID 15994231
- [Result] Park SG, Ryu HM, Lim SO, Kim YI, Hwang SB, Jung G. Interferon-gamma inhibits hepatitis B virus-induced NF-kappaB activation through nuclear localization of NF-kappaB-inducing kinase. Gastroenterology. 2005 Jun;128(7):2042-53. doi: 10.1053/j.gastro.2005.03.002. PMID 15940636
- [Result] Bissett J, Eisenberg M, Gregory P, Robinson WS, Merigan TC. Recombinant fibroblast interferon and immune interferon for treating chronic hepatitis B virus infection: patients' tolerance and the effect on viral markers. J Infect Dis. 1988 May;157(5):1076-80. doi: 10.1093/infdis/157.5.1076. No abstract available. PMID 3129521
- [Result] Porres JC, Mora I, Gutiez J, Bartolome J, Quiroga JA, Bas C, Compernolle C, Ordi J, Chocarro A, Carreno V. Antiviral effect of recombinant gamma interferon in chronic hepatitis B virus infection: a pilot study. Hepatogastroenterology. 1988 Feb;35(1):5-9. PMID 2452123
- [Result] Di Bisceglie AM, Rustgi VK, Kassianides C, Lisker-Melman M, Park Y, Waggoner JG, Hoofnagle JH. Therapy of chronic hepatitis B with recombinant human alpha and gamma interferon. Hepatology. 1990 Feb;11(2):266-70. doi: 10.1002/hep.1840110217. PMID 2106474
- See also: Huntington Medical Research Institutes — http://www.hmri.org/
- See also: Myron J. Tong, PhD, MD — http://www.uclahealth.org/body.cfm?xyzpdqabc=0&id=479&action=detail&ref=20715